CLINICAL TRIAL: NCT04815278
Title: NC Works4Health: Reducing Chronic Disease Risks in Socioeconomically Disadvantaged, Unemployed Populations
Acronym: NCW4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 21-0859; 1R01MD012832-01A1 (NIH)
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Chronic Disease; Psychological Distress
Keywords: Unemployment; Weight Maintenance; Unintentional Bias; Employment Services; Self-Monitoring; Perceived Workplace Support; Step Count; Coping Strategies; Blood Pressure; Food Tracking; Problem-Solving; Weight Loss; Underemployment
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease; Weight Loss | interventions — Occupations

STUDY DESIGN:
Intervention Model Description: Random 2x2 factorial design. The temporal nature of the phenomenon under study requires individuals (DSS-E participants) are first randomized to the individual-level treatment group, follow them as they are naturally hired into employment settings, and then enroll / randomize / allocate employers to the employer-level treatment group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Experimental): Participants will receive usual DSS employment services that include, but are not limited to, consultation with an employments specialist, resume writing guidance, educational classes and attendance at job fairs. Participants will have access to a delayed, attenuated online-only version of the CDPP at the time they complete the 12 month data collection. This version will provide all modules, self-monitoring options (including through use of a Fitbit contingent on the completion of the 12 month data collection) but will not include face-to-face or phone lifestyle coach sessions.
  Interventions: Behavioral: Delayed, attenuated Chronic Disease Prevention Program (CDPP)
- Employer Intervention Only (Experimental): Participants will receive usual DSS employment services and an employer level workplace equity, job & health supports intervention. The employer intervention will include an implicit bias workshop and supervisor support training in addition to regular supervisor check-ins every other week.
  Interventions: Behavioral: Workplace Equity, Job and Health Supports Employer Intervention
- CDPP Only (Experimental): Participants will receive the individual level CDPP intervention and no employer intervention. The CDPP is a 24-week online curriculum that consists of 8 learning modules and 7 lifestyle coach sessions. Content for the program will include healthy lifestyle habits, managing stress and staying motivated.
  Interventions: Behavioral: Immediate Chronic Disease Prevention Program (CDPP)
- CDPP and Employer Intervention (Experimental): Participants will receive the individual level CDPP intervention and employer level workplace equity, job & health supports intervention. The CDPP is a 24-week online curriculum that consists of 8 learning modules and 7 lifestyle coach sessions and check-ins. Content for the program will include healthy lifestyle habits, managing stress and staying motivated. The employer intervention will include an implicit bias workshop and supervisor support training, in addition to regular supervisor check-ins every other week..
  Interventions: Behavioral: Immediate Chronic Disease Prevention Program (CDPP); Behavioral: Workplace Equity, Job and Health Supports Employer Intervention

INTERVENTIONS:
Behavioral: Immediate Chronic Disease Prevention Program (CDPP) — The CDPP is an adaptation of the Diabetes Prevention Program (DPP). It will take place over a 24 week period and involve online instruction and individualized lifestyle coaching sessions. The online classroom curriculum includes 8 modules: Goal setting, self-monitoring and problem solving (M1), Managing stress and negative thoughts (M2), Healthy eating (M3), Taking more steps (M4), Keeping alcohol in check (M5), Lifestyle change (M6), Taking charge of what (and who) is around you (M7), and Staying motivated (M8). The lifestyle coaches will meet in person and over the phone intermittently over the 24 week period (Weeks 2, 4, 6, 10, 12, 16, 24).
  Arms: CDPP Only; CDPP and Employer Intervention
Behavioral: Workplace Equity, Job and Health Supports Employer Intervention — The employer intervention combines implicit bias awareness training for supervisors of hired DSS-E clients, and regular, structured, interactions between supervisors and DSS-E hires.
  Arms: CDPP and Employer Intervention; Employer Intervention Only
Behavioral: Delayed, attenuated Chronic Disease Prevention Program (CDPP) — Participants will have access to a delayed, attenuated online-only version of the CDPP at the time they complete the 12 month data collection. This version will provide all modules, self-monitoring options (including through use of a Fitbit contingent on the completion of the 12 month data collection) but will not include face-to-face or phone lifestyle coach sessions.
  Arms: Control Group

SUMMARY:
The proposed study, NC Works4Health (NCW4H), builds on the strengths of long-standing academic-community research partnerships between this UNC at Chapel Hill (UNC) team of investigators and key stakeholders across health, social service, employment, and economic development sectors. The overall goal of this study is to test the effectiveness of a multilevel intervention that can be readily adopted by communities to reduce chronic disease risks in socioeconomically disadvantaged populations by (a) embedding prevention efforts in DSS-E programs at the individual level, and (b) enhancing supervisor supports for DSS-E hires at the employer level. Interventions at each level, and their joint effects, are designed to mitigate the psychological, behavioral, and clinically relevant risks for chronic disease onset, morbidity, and comorbidity that accrue with unemployment and the employment-entry transition.

DETAILED DESCRIPTION:
Studies have shown that a single episode of unemployment can trigger a cascade of stress-related coping and behavioral processes that have deleterious effects on health. Notably, this cascade not only frequently results in psychological distress, but also accelerated weight gain (persisting up to 10 years regardless of re-employment), and elevated blood pressure. As such, individuals who experience unemployment are at a much higher risk for chronic disease development, comorbidity, and early mortality. Given inequities in the labor market, socioeconomically disadvantaged groups (i.e., those with less education, less income or wealth, and/or who are racial/ethnic minorities) are disproportionately, and more adversely affected by both unemployment and chronic disease, and feel this burden acutely in their everyday lives. Socioeconomically disadvantaged adults often receive public assistance benefits during unemployment episodes as well as job training and placement services through Department of Social Services Employment (DSS-E) programs; however, these programs do not include prevention-focused content to reduce the chronic disease risks that accrue during unemployment episodes. In addition, DSS-E efforts to help individuals succeed in securing and performing in a new job are often thwarted by implicit 'welfare'-related bias and insufficient supports in workplaces into which DSS-E clients are hired. Although the current absence of chronic disease prevention in DSS-E programs and lack of supports for DSS-E hires in workplaces compound chronic disease risks, it is also an area in which communities can address social determinants that are known to produce health inequities.

The proposed study, NC Works4Health (NCW4H), builds on the strengths of long-standing academic-community research partnerships between this UNC at Chapel Hill (UNC) team of investigators and key stakeholders across health, social service, employment, and economic development sectors. The overall goal of this study is to test the effectiveness of a multilevel intervention that can be readily adopted by communities to reduce chronic disease risks in socioeconomically disadvantaged populations by (a) embedding prevention efforts in DSS-E programs at the individual level, and (b) enhancing supervisor supports for DSS-E hires at the employer level. Interventions at each level, and their joint effects, are designed to mitigate the psychological, behavioral, and clinically relevant risks for chronic disease onset, morbidity, and comorbidity that accrue with unemployment and the employment-entry transition. By collaborating across sectors to reduce health inequities, the specific aims will be met in two phases:

Phase I

With community partners and key stakeholders, make minor adaptations to two evidence-based interventions for use in a multilevel intervention that incorporates: (a) a chronic disease prevention program (CDPP) (individual level)into current DSS-E programs for unemployed adults, and (b) supervisor support in the workplace (employer level)into an existing network of employers with jobs that match the skill set of the DSS-E program population.

Phase II

Aim 1. To test the main effects of (a) the individual-level NC Works4Health intervention (Usual DSS-E + CDPP) compared to Usual DSS-E Support, and (b) the employer-level NC Works4Health intervention compared to usual workplace supports on primary and secondary outcomes, over time (at 3, 6, and 12 months from baseline), using a randomized, 2x2 factorial design.

Aim 2. To test the joint effect of the individual-level + employer-level NC Works4Health interventions on primary and secondary outcomes, over time (at 3, 6, and 12 months from baseline).

In the primary outcomes, the investigators expect to see a decrease in psychological distress, weight gain, and blood pressure in groups receiving the intervention at each level, with the greatest decreases in the outcomes observed in the group receiving both the individual- and employer-level interventions.

Secondary outcomes include situational stress, coping style, health behaviors, perceived workplace support, health-related employment functioning and employment duration.

ELIGIBILITY:
Inclusion Criteria:

* receiving DSS-E services
* between the age of 18 and 64 years old
* unemployed
* fluent and able to read English

Exclusion Criteria:

* receiving or applied for disability benefits
* pregnant
* Any of the following chronic conditions: severe high blood pressure (with a reading of 180/110 or higher in the past 6 months), a health condition or injury that has left you unsteady, or unbalanced when you walk, a history of falling in the past 6 months, cancer that is actively being treated with chemotherapy of radiation to your chest or abdomen (stomach area), inflammatory bowel disease (such as Crohn's disease, or ulcerative colitis), an implanted cardiac defibrillator (a small device placed under the skin on your chest to help your heart function)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 455 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Mean Psychological Distress Scores at Baseline | Baseline (Month 0)
  The Patient Health Questionnaire (PHQ-8) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It is an 8 item scale with each item rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of depression while lower scores indicate lower levels of depression. Scores range from 0-24.
  The Generalized Anxiety Disorder (GAD-7) is a 7 item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Items are rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of anxiety while lower scores indicate lower levels of anxiety. Scores range from 0-21.
  To obtain an aggregate score for Psychological Distress, the PHQ & GAD will be combined. Scores will range from 0-45.
Mean Psychological Distress Scores at Month 3 | 3 Months
  The Patient Health Questionnaire (PHQ-8) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It is an 8 item scale with each item rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of depression while lower scores indicate lower levels of depression. Scores range from 0-24.
  The Generalized Anxiety Disorder (GAD-7) is a 7 item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Items are rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of anxiety while lower scores indicate lower levels of anxiety. Scores range from 0-21.
  To obtain an aggregate score for Psychological Distress, the PHQ & GAD will be combined. Scores will range from 0-45.
Mean Psychological Distress Scores at Month 6 | Month 6
  The Patient Health Questionnaire (PHQ-8) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It is an 8 item scale with each item rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of depression while lower scores indicate lower levels of depression. Scores range from 0-24.
  The Generalized Anxiety Disorder (GAD-7) is a 7 item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Items are rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of anxiety while lower scores indicate lower levels of anxiety. Scores range from 0-21.
  To obtain an aggregate score for Psychological Distress, the PHQ & GAD will be combined. Scores will range from 0-45.
Mean Psychological Distress Scores at Month 12 | Month 12
  The Patient Health Questionnaire (PHQ-8) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It is an 8 item scale with each item rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of depression while lower scores indicate lower levels of depression. Scores range from 0-24.
  The Generalized Anxiety Disorder (GAD-7) is a 7 item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Items are rated on a 4 point scale from "Not at all" (score 0) to "Nearly every day" (score 3). Higher scores indicate higher levels of anxiety while lower scores indicate lower levels of anxiety. Scores range from 0-21.
  To obtain an aggregate score for Psychological Distress, the PHQ & GAD will be combined. Scores will range from 0-45.
Weight at Baseline | Baseline (Month 0)
  Weight will be measured using the Tanita WB-800 Plus professional grade scale. Lightweight and portable, it has a weight capacity of 660 lbs, and has been used in studies of weight gain prevention by others on the research team.
Weight at Month 3 | Month 3
  Weight will be measured using the Tanita WB-800 Plus professional grade scale. Lightweight and portable, it has a weight capacity of 660 lbs, and has been used in studies of weight gain prevention by others on the research team.
Weight at Month 6 | Month 6
  Weight will be measured using the Tanita WB-800 Plus professional grade scale. Lightweight and portable, it has a weight capacity of 660 lbs, and has been used in studies of weight gain prevention by others on the research team.
Weight at Month 12 | Month12
  Weight will be measured using the Tanita WB-800 Plus professional grade scale. Lightweight and portable, it has a weight capacity of 660 lbs, and has been used in studies of weight gain prevention by others on the research team.
Blood Pressure at Baseline | Baseline (Month 0)
  Blood Pressure will be assessed using the American Heart Association Guidelines for BP measurement and the Omron HEM-705CPN, which meets strict calibration standards and is validated at +/- 3-5 mmHg (millimeters of mercury).
Blood Pressure at Month 3 | Month 3
  Blood Pressure will be assessed using the American Heart Association Guidelines for BP measurement and the Omron HEM-705CPN, which meets strict calibration standards and is validated at +/- 3-5 mmHg (millimeters of mercury).
Blood Pressure at Month 6 | Month 6
  Blood Pressure will be assessed using the American Heart Association Guidelines for BP measurement and the Omron HEM-705CPN, which meets strict calibration standards and is validated at +/- 3-5 mmHg (millimeters of mercury).
Blood Pressure at Month 12 | Month 12
  Blood Pressure will be assessed using the American Heart Association Guidelines for BP measurement and the Omron HEM-705CPN, which meets strict calibration standards and is validated at +/- 3-5 mmHg (millimeters of mercury).

SECONDARY OUTCOMES:
Scores on Situational Stress Scale | Up to 12 months
  Situational stress will be measured by the Perceived Stress Scale (PSS), a 14 item measure of the extent to which the circumstances of one's life are appraised as stressful. Each item is rated on a 5-point scale from "Never" (score 0) to "Very Often" (score 4). Higher scores indicate higher levels of stress while lower scores indicate lower levels of stress. Scores range from 0-56. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Scores on Coping Strategies Scale | Up to 12 months
  Coping style will be measured by the Coping Strategies Inventory (CSI), a 32 item measure designed to assess coping thoughts and behaviors in response to a specific stressor. Each item is rated on a 5-point scale from "Not at All" (score 1) to "Very Much" (score 5). Higher scores indicate higher levels of coping while lower scores indicate lower levels of coping. Scores range from 32-160. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Scores on Health Self-Regulation Scale | Up to 12 months
  Health Self-Regulation will be gauged by the Index of Self-Regulation (ISR) which measures Stimulus Control, Reconditioning, and Behavioral Monitoring self-regulation domains. The ISR is a 12- item measure rated on a 6-point scale from "Strongly Disagree" (score 1) to "Strongly Agree" (score 6). Higher scores indicate higher levels of self-regulation while lower scores indicate lower levels of self-regulation. Scores range from 12-72. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Number of Steps Taken as Determined by ActiGraph Accelerometer | Up to 12 months
  ActiGraph wGT3X-BT, 3-axis accelerometers will measure physical activity over 3 days. These are small, water resistant, lightweight, and worn on the wrist or hip. Data download electronically; algorithm generates mean number of steps taken. Measurements will be assessed for a 3 day period at Baseline (Month 0), and Months 3, 6, and 12.
Physical Activity Intensity as Determined by ActiGraph Accelerometer | Up to 12 months
  ActiGraph wGT3X-BT, 3-axis accelerometers will measure physical activity over 3 days. These are small, water resistant, lightweight, and worn on the wrist or hip. Data download electronically; algorithm generates mean physical activity intensity values using using units of Moderate to Vigorous Physical Activity (MVPA). Measurements will be assessed for a 3 day period at Baseline (Month 0), and Months 3, 6, and 12.
Sedentary Bouts as Determined by ActiGraph Accelerometer | Up to 12 months
  ActiGraph wGT3X-BT, 3-axis accelerometers will measure physical activity over 3 days. These are small, water resistant, lightweight, and worn on the wrist or hip. Data download electronically; algorithm generates sedentary "bouts" in units of time (seconds). Measurements will be assessed for a 3 day period at Baseline (Month 0), and Months 3, 6, and 12.
MET Rate as Determined by ActiGraph Accelerometer | Up to 12 months
  ActiGraph wGT3X-BT, 3-axis accelerometers will measure Metabolic Equivalent (MET) physical activity over 3 days. These are small, water resistant, lightweight, and worn on the wrist or hip. Data download electronically; algorithm generates a mean MET rate. Measurements will be assessed for a 3 day period at Baseline (Month 0), and Months 3, 6, and 12.
Dietary Intake Log | Up to 12 months
  NCI's Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24®) will collect all dietary intake data over 3 days. With portion size images, accuracy of the ASA24® (+/- 3.7g) now supersedes that of the long-standing gold standard. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Scores on Alcohol Use Scale | Up to 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Alcohol Use scale will assess the consumption quantity and frequency, and problem drinking. It is a 14 item measure rated on a 5-point scale from "Never" (score 1) to "Almost Always" (score 5). Higher scores indicate higher levels of alcohol use while lower scores indicate lower levels of alcohol use. Scores range from 14-70. Outcome data will be collected at Baseline (Month 0) and a Months 3, 6, and 12.
Scores on Smoking Quantity Scale | Up to 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Smoking Module assesses smoking quantity. The PROMIS Smoking module is a 10 item measure rated on a 5-point scale from "Never" (score 1) to "Always" (score 5). Higher scores indicate higher levels of smoking while lower scores indicate lower levels of smoking. Scores range from 10-50. These scores will only be reported for participants that indicate they are current smokers. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Responses to Motivation to Stop Smoking | Up to 12 months
  The Motivation to Stop Scale (MTSS) assesses readiness to quit. The MTSS is a 1 item multiple choice measure with 7 options. These scores will only be reported for participants that indicate they are current smokers. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Scores on Employment Functioning Scale | Up to 12 months
  The Work Limitations Questionnaire (WLQ) captures health-related absenteeism and presenteeism. The WLQ is a 25 item measure rated on a 5-point scale from "None of the time" (score 1) to "All of the time" (score 5). Higher scores indicate higher levels of employment functioning while lower scores indicate lower levels of employment functioning. Average item scores will be calculated to a 25-125 range. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Mean Change in Perceived Discrimination Scores | Up to 12 Months
  The Perceived Supervisor Discrimination scale (adapted) is an aggregate measure of two short measures: the job harassment index and the treated unfairly on job index. The job harassment index consists of 2 items and the treated unfairly on job index consists of 3 items. Each is rated on the same 5 point scale from Never (score 0) to 1+ times a week (score 4). Higher scores indicate higher occurrences of harassment/unfair treatment. Scores range from 0-20. Because the 2 sub-scales are rated on the same 5-point scale, the scores will be added together for an aggregate score. Measurements will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Mean Change in Perceived Supervisor Support Scores | Up to 12 Months
  The Perceived Supervisor Support Scale is a 12 item measure that quantitatively captures employee's relationship with their supervisor and the extent to which they believe their supervisor is supportive of them. The scale is adapted from the Perceived Organizational Support scale by replacing the word "Organization" with "Supervisor. Respondents indicate their agreement with each item using a 7-point Likert-type scale (0=strongly disagree, 6=strongly agree). Higher scores indicate higher levels of agreement. Scores range from 0-72. Measurements will be assessed at Baseline (Month 0), and Months 3, 6, and 12.
Proportion of Days Employed | Up to 12 months
  Employment duration will be measured by Person-Time Employed (proportion of days employed regardless of breaks in employment) over the entire one year study period. Employment start and stop dates will be collected at each of the data collection time points (Baseline (Month 0), and Months 3, 6, and 12). Employment duration proportion will be calculated after the 12 month data collection.
Weeks of Continuous Employment | Up to 12 months
  Employment duration will be measured by Continuous Employment (number of consecutive weeks employed, with any reported work in a given week counted as a positive week of employment) over the entire study period. Continuous weeks of employment will be collected at each of the data collection time points (Baseline (Month 0), and Months 3, 6, and 12). Weeks continuous employment will be calculated after the 12 month data collection.
Number of Times of Healthcare Utilization | Up to 12 months
  Participants will self-report their health care utilization by point of service in the previous three months (e.g., ER visits, meds). Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Total Amount of Supplementary Out-of-pocket costs | Up to 12 months
  Participants will self-report total amount of supplementary out-of-pocket costs (e.g., dietary supplements, gym classes, health-related equipment) in the previous three months. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Scores on Organizational Citizenship Behaviors Checklist | Up to 12 months
  The Organizational Citizenship Behaviors Checklist (OCB-C) Scale assesses the frequency of employee behaviors that go above and beyond job responsibilities. The OCB-C is a 20-item scale that is scored on a 5-point Likert scale (1= Never, 5= Every day). High scores indicate more organizational citizenship behaviors. Low scores indicate less organizational citizenship behaviors. Scores range from 20-100. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Scores on General Health | Up to 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health assesses general health. The PROMIS Global Health module is a 10 item measure rated on a 5-point scale from "Excellent" (score 1) to "Poor" (score 5). Higher scores indicate poorer health while lower scores indicate better health. Scores range from 10-50. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Health Care Provider Status | Up to 12 months
  Participants will answer a single item that asks if they currently have a primary health care provider. Answer choices are binary; yes or no. This item will not be scored. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Chronic Conditions | At Baseline (Month 0)
  Participants will answer a single item that asks for all chronic conditions they have ever had that have been diagnosed by a health care professional. There is a list of 28 chronic condition options. Participants may choose multiple conditions. This item will not be scored.
Health Management Apps/Programs/Wearables Use | Up to 12 months
  The Health Management Use scale measures how frequently participants have used apps, gadgets, or strategies to manage their health in the last 3 months. It is a 13 item measure rated on a 4-point scale from "Used daily or almost daily" (score 1) to "Have not used" (score 4) scale. Higher scores indicate less health management use while lower scores indicate more health management use. Scores range from 13-52. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Medication Covariates | Up to 12 months
  A single item about current medications: Diabetes (Thiazolidinediones, Sulfonylureas, insulin), Anti-psychotics (Haloperidol,Clozapine, Risperidone, Olanzapine, Quetiapine, Lithium, Valproic acid, Carbamezapine), Anti-depressants (Amitriptyline, Imipramine, Paroxetine, Escitalopram, Citalopram, Mirtazapine, Sertraline), Anti-epileptics (Valproate, Divalproex, Carbamazepine, Gabapentin, nortriptyline, valproic acid), Steroids (Prednisone, prednisolone, Cortisone, methylprednisolone, Anti-hypertensives, Propranolol, Metoprolol, Amiodipine, Conidine, atenolol), Diabetes (Metformin, Liraglutide), Bronchodilator (Theophylline), Stimulants (Methylphenidate, Dextroamphetamine), Anticonvulsant (Topiramate), Antidepressant (Bupropion, Fluoxetine), Anti-inflammatory (Sulphasalazine), Other weight loss medications (Orlistat, Lorcaserin, Phentermine-topiramate, Naltrexone-bupropion). The item is multiple choice. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.

OTHER OUTCOMES:
Responses to CDC Scorecard | Up to 60 months
  The Center for Disease Control and Prevention (CDC) ScoreCard consists of 154 yes or no binary questions that measure worksite health strategies in 16 areas being implemented in employer organizations. It will be used to assess and adjust for (if necessary) employer group equivalence, and for guiding generalizing findings to a broader population of employers. Outcome data will be collected at Baseline (Month 0) and every 12 months.
Scores on Chronic Financial Strain Scale | Up to 12 months
  The Chronic Financial Strain (CFS) scale (5 items) assesses the frequency that funds are unavailable to purchase basic necessities (i.e., food, medical care, clothing). Items are rated on a 5-point scale from "Never" (score 0) to "Always" (score 4). Lower scores indicate lower levels of financial strain while higher scores indicate higher levels of financial strain. Scores range from 0-20. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.
Scores on Effort-Reward Imbalance Scale | Up to 12 months
  The Effort-Reward Imbalance-Short (ERI-S) scale (16 items) will measure work effort, reward, and commitment. Item responses are scored on a 4-point Likert-type scale (1 = strongly disagree, 4 = strongly agree). High scores indicate high effort and high reward. Scores range from 16-64. Outcome data will be collected at Baseline (Month 0), and Months 3, 6, and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Kneipp, Ph. D, Principal Investigator — UNC School of Nursing
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, UNC will prepare a final, de-identified limited-access dataset suitable for sharing with other researchers that will be made available 9-36 months following publication. UNC has had considerable experience with producing deidentified datasets, because it has prepared them for a number of the studies it is coordinating or has coordinated. De-identification will include removal of obvious identifiers such as names and addresses. It will also include examination of less obvious potentially identifying variables. Continuous variables with extreme values may have the extremes truncated. Height and weight are examples of such variables. Categorical variables with small numbers of participants in some categories may have these categories pooled with larger categories.
Supporting Information: Study Protocol
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Access Criteria: The limited-access dataset will be made available at the end of the study. Data will be released in a .csv file. Researchers wishing to use the dataset will be required to obtain approval from UNC using an agreement form that clearly specifies the intended analyses as well as assurances that HIPAA regulations will be followed. If approval is granted, the dataset will be supplied on a CD, or shared using a secure, password-protected medium. It will also include documentation describing the variables in the dataset and copies of the data collection forms used to collect the data.

DOCUMENTS (1):
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04815278/ICF_000.pdf